CLINICAL TRIAL: NCT05140187
Title: Adoptive Immunotherapy With Donor-derived CMV-TCR-T Cells for Patients With CMV Infection After Allogenic HSCT
Brief Title: CMV-TCR-T Cells for CMV Infection After Allogenic HSCT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2021-344-01
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: CMV Infection After Allogenic HSCT
Keywords: CMV; HSCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMV-TCR-T cells (Experimental): The patients with CMV infection after HSCT will receive one to three infusions of donor-derived CMV-TCR-T cells, with the escalated dose ranging from 1×10^3/kg to 5×10^5/kg CMV-TCR-T cells per dose.
  Interventions: Biological: CMV-TCR-T cells

INTERVENTIONS:
Biological: CMV-TCR-T cells — The patients with CMV infection after HSCT will receive one to three doses of donor-derived CMV-TCR-T cells, with the escalated doses including 1×10^3/kg, 1×10^5/kg, and 5×10^5/kg CMV-TCR-T cells per dose.

SUMMARY:
This is a multi-center, single arm, open-label, phase I study to determine the safety and effectiveness of CMV-TCR-T cell immunotherapy in treating CMV virus infection after allogenic HSCT.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) infection after allogeneic hematopoietic stem cell transplantation (HSCT) is common and can be lethal without prompt treatment. In this prospective study, HLA-A*02:01/11:01/24:02-restricted CMV-specific T cell receptor (TCR) will be introduced into the T cells of HSCT donors by ex vivo lentiviral transduction to generate CMV-TCR-T cells. An escalated dose ranging from 1×10^3/kg to 5×10^5/kg of CMV-TCR-T cells will be infused into patients with CMV infection. The safety, efficacy, pharmacokinetics and cytokine levels of allogenic CMV-TCR-T cell therapy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-60 years, gender unlimited.
2. Diagnosed with hematologic malignancies and have undergone allogeneic hematopoietic stem cell transplantation (allo-HSCT), with CMV infection after allo-HSCT.
3. Karnofsky Score ≥ 70 or Lansky Score ≥ 50.
4. TCR-T cell donor inclusion criteria:

1) Age ≥ 8 years; 2) Understand and voluntarily sign informed consent and are willing to comply with laboratory tests and other research procedures; 3) ≥ 3/6 HLA match with TCR-T cell recipients enrolled; 4) Lymphocyte count = (0.8~4) × 10^9/L; 5) Have sufficient venous circulation, without any symptoms that do not allow blood cell isolation.

Exclusion Criteria:

1. Patients with active aGVHD one day before TCR-T cell infusion.
2. Patients with severe kidney disease (Cr > 3×normal value), liver damage (TBIL >2.5×upper limit of normal value, ALT and AST > 3×upper limit of normal value) or heart failure (NYHA heart function grade IV) one week before TCR-T cell infusion.
3. Anticipated to take immunosuppressive hormones on the day of TCR-T cell infusion.
4. Have other malignancies.
5. Have relapsed and uncontrolled hematologic malignancies.
6. Serologically positive for HIV-Ab or TAP-ab.
7. Pregnant or lactating women.
8. Anticipated to have other cell therapies in 4 week post TCR-T cell infusion.
9. Participated in any other clinical study of drugs and medical devices before 30 days of enrollment.

11. Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.

12. TCR-T cell donor exclusion criteria:

1. Positive for any of the following: HbsAg, HBeAg, HBV-DNA, HCV-Ab, HCV-RNA, HIV-Ab, TP-Ab, EBV-DNA or CMV-DNA;
2. Other uncontrolled infection;
3. Have taken immunosuppressive drugs 1 week before PBMC collection;
4. Any condition that would, in the investigator's judgment, make it unsuitable for the donors to be enrolled.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 year
  Percentage of participants with adverse events.

SECONDARY OUTCOMES:
Changes of CMV-DNA copies number | 1 year
  Quantitative PCR will be used to determine viral copy numbers in peripheral blood.
Persistence of CMV-TCR-T cells | 1 year
  Quantitative PCR using primers specific for the gene encoding CMV-TCR will be used to determine the number of circulating CMV-TCR-T cells in peripheral blood post infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ma C, Chen P, Du J, Wang L, Lu N, Sun J, Qilong X, Wang Y, Dou L, Liu DH. Adoptive transfer of CMV-specific TCR-T cells for the treatment of CMV infection after haploidentical hematopoietic stem cell transplantation. J Immunother Cancer. 2024 Jan 6;12(1):e007735. doi: 10.1136/jitc-2023-007735. PMID 38184303